CLINICAL TRIAL: NCT01130766
Title: Randomized Phase III Trial of Stereotactic Radiosurgery (SRS) Versus Observation for Patients With Asymptomatic Cerebral Oligo-metastases in Non-small Cell Lung Cancer (NSCLC)
Brief Title: Asymptomatic Brain Metastasis in Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myungju Ahn Ph.D., M.D., Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-01-059
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Asymptomatic brain metastasis; Stereotactic radiosurgery (SRS)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stereotactic radiosurgery (SRS) (Experimental)
  Interventions: Procedure: stereotactic radiosurgery (SRS)
- observation (No Intervention)

INTERVENTIONS:
Procedure: stereotactic radiosurgery (SRS) — Stereotactic radiosurgery using γ-rays from radioactive Cobalt-60 installed in Gamma Knife (Elekta Instruments, Stockholm, Sweden)
  Arms: stereotactic radiosurgery (SRS)

SUMMARY:
The prognosis of NSCLC patients with asymptomatic brain metastasis, who are not treated with SRS or WBRT has not been fully investigated yet. This randomized phase III trial is conducted to determine the exact role of SRS in NSCLC patients with asymptomatic oligo brain metastases whether early treatment with SRS would improve survival even in patients with asymptomatic brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer with synchronous brain metastases (diagnosis of brain lesion before or within 2 months from diagnosis of the primary site tumor)

  * One to 4 intraparenchymal brain metastases by contrast-enhanced MRI, meeting the following criteria:

    1. Well circumscribed tumor(s) with brain edema Grade 0-1
    2. Maximum diameter ≤ 3.0 cm

       * No prior complete resection of all known brain metastases or RT ④ No leptomeningeal metastases by MRI or cerebrospinal fluid evaluation

         * Patients without any symptoms or signs from brain metastases (RTOG neurologic functions status of 0) ⑥ Age, 18 and over ⑦ ECOG performance status 0-1 ⑧ Written informed consent

       Exclusion Criteria:
* severe co-morbid illness and/or active infections ② pregnant or lactating women

  * RTOG neurologic function status of 1~4 ④ Uncontrollable extracranial metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months

SECONDARY OUTCOMES:
time to CNS progression | 36 months
time to symptomatic brain metastasis | 36 months
quality of life | 36 months
cause of death (neurologic vs. others) | 36 months
neurocognitive function | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Myungju Ahn, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea